CLINICAL TRIAL: NCT05719402
Title: Quantitative Assessment of Intestinal Motility on Bowel Ultrasound in Patients With Inflammatory Bowel Disease: a Feasibility, Observational, Prospective, Monocentric Study
Brief Title: Quantitative Assessment of Intestinal Motility on Bowel Ultrasound in Patients With Inflammatory Bowel Disease: a Feasibility, Observational, Cross-sectional, Monocentric Study
Acronym: MOTUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, MARIANGELA ALLOCCA, Gastroenterologist, IRCCS San Raffaele
Other Study IDs: MOTUS
Record Dates: First submitted 2023-01-27; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: non-interventional prospective cross-sectional observational study — to investigate the feasibility of using intestinal motility quantified by intestinal ultrasound (US) to evaluate disease activity. The outcomes of intestinal motility detected by ultrasound will be compared with endoscopic and histopathological reference standards in adult patients with IBD

SUMMARY:
Inflammatory bowel diseases (IBD), such as ulcerative colitis (UC) and Crohn's disease (CD), are chronic, relapsing and destructive inflammatory disorder of the intestinal wall. A treat-to-target approach with tight monitoring of intestinal inflammatory lesions is recommended to prevent organ damage and impaired quality of life. Because clinical scores and laboratory assessments have shown poor correlation with intestinal inflammation, endoscopic investigation has to be performed frequently as a reference standard. Due to the fact that colonoscopy (CS) is poorly accepted by patients, expensive, time consuming and harbors the risk of complications, new imaging strategies are required to overcome invasive procedures. The aim of this non-interventional prospective cross-sectional observational study is to investigate the feasibility of using intestinal motility quantified by intestinal ultrasound (US) to evaluate disease activity. The outcomes of intestinal motility detected by ultrasound will be compared with endoscopic and histopathological reference standards in adult patients with IBD

DETAILED DESCRIPTION:
This is a feasibility, observational, cross-sectional, monocentric study on the evaluation of a non-invasive US approach based on the intestinal motility detection for the assessment of activity in IBD.

About 100 IBD patients under treatment at the Gastroenterology Department of the San Raffaele Hospital will be enrolled between September 2022 and September 2023. According to the observational nature of the study, all the visits and procedures described below will be performed according to the diagnostic and therapeutic assignment required by clinical practice for the patients under study. The choice of treatment will be made by the referring physicians according to the international ECCO guidelines. Therefore, the choice of assigning the patient to the diagnostic and therapeutic procedures deemed most appropriate for each case is completely independent of the study.

IBD patients will be prospectively identified and consecutively recruited. Within 7 days from the colonoscopy, patients will undergo complete clinical assessment. Harvey-Bradshaw Index (HBI) and partial Mayo score (PMS) will be calculated in Crohn's disease and in ulcerative colitis, respectively. Blood and stool samples will be obtained for C-reactive protein (CRP) and fecal calprotectin (FC) measurements.

Bowel US will be performed, in a blinded fashion, after 6-8 hour fasting, using an Aloka Arietta 750 with convex (5-1 MHz) and microconvex probes (4-8 MHz), by two expert gastroenterologists of the IBD center. Neither preparation nor contrast will be used. anonymized cineloops of the ileum segment and sigmoid colon in CD and sigmoid colon in UC, will be recorded and sent to an external cloud platform Entrolytics which is a PACS for ultrasound, for the assessment of motility through a specific software.

Any treatment will be kept stable in the interval between the two procedures. The informations obtained on the analysis of intestinal motility will not be used for therapeutic purposes on patients who will follow the therapeutic path provided by the ECCO reference guidelines.

For this reason motility analysis will not be used for clinical purposes, but for research purposes only.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* established diagnosis since at least 3 months requiring colonoscopy, US and histologic evaluation of tissue biopsies according to ECCO international guidelines 3-5
* 50 CD ileo-colonic patients, 25 in endoscopic activity (as defined by a SES-CD > 2), 25 in endoscopic remission (as defined by a SES-CD < 2), independently from treatment;
* 50 UC patients, 25 in endoscopic activity (as defined by a Mayo endoscopic score > 2), 25 in endoscopic remission (as defined by a Mayo endoscopic score < 2), independently from treatment.

Exclusion Criteria:

* Patients with inflammation restricted to the rectum (≤ 15 cm from the anal verge);
* UC patients without involvement of sigmoid colon or inability to reach the sigmoid colon by CS;
* CD patients without ileal involvement or inability to reach the ileum by CS;
* Patients with severe UC (defined as a Mayo global score > 12, requiring hospitalization);
* Pregnancy;
* Previous intestinal surgery;
* Concomitant intestinal infection (e.g. Clostridium difficile);
* Cirrhosis or intra-abdominal ascites.
* Patients not able to comply with any study procedure;
* Patients not able to understand and give informed consent form;
* Patients with any contraindication to any study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 adult IBD patients (established diagnosis since at least 3months) at the Gastroenterology Department of the San Raffaele Hospital requiring colonoscopy, US and histologic evaluation of tissue biopsies according to ECCO international guidelines
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-11-25 (Estimated); Study Completion 2024-11-25 (Estimated)

PRIMARY OUTCOMES:
outcomes of intestinal motility detected by ultrasound will be compared with endoscopic and histopathological reference standards in adult patients with IBD. | 1 DAY
  outcomes of intestinal motility detected by ultrasound will be compared with endoscopic and histopathological reference standards in adult patients with IBD.

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Allocca, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Mariangela Allocca, Milan, Italy